CLINICAL TRIAL: NCT07336914
Title: Effect of Conventional vs Intensive Management on Gestational Diabetes and Maternal Fetal Outcomes: Randomized Controlled Trial.
Brief Title: Effect of Conventional vs Intensive Management on Gestational Diabetes and Maternal Fetal Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Northwest General Hospital and Research centre (Network); Hayatabad Medical Complex (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/09
Record Dates: First submitted 2025-12-10; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes Mellitus (GDM); Intensive Management; Randomized Controlled Trial (RCT); Glycemic Control; Maternal Health
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups (arms), and each group receives a different intervention concurrently.
Masking Description: The nature of the interventions (monthly vs. weekly follow-up, different monitoring intensities) makes blinding of participants and care providers impossible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Management Group (Active Comparator): This group receives standard care for conventional management of GDM identified via survey in government and private sectors. This includes monthly follow-up visits with basic lifestyle modification and counselling on dietary and physical acitivity assessed via questionnaires (PDAQ and PPAQ). Medication (insulin or oral agents like metformin) is only introduced if glycemic targets are not achieved through lifestyle modifications alone. Blood glucose monitoring is performed at a standard frequency (e.g., pre- and post-meal).
  Interventions: Other: Usual care
- Intensive Management Group (Experimental): This group receives a standardized, intensive multidisciplinary intervention. It includes weekly telephonic monitoring, personalized low-carbohydrate/calorie diet plans, and structured moderate and intense exercise based on their activty level. Pharmacotherapy (insulin, metformin, etc.) is initiated proactively if glucose levels are not controlled within two weeks. Enhanced fetal monitoring via frequent ultrasounds is also included to assess growth and amniotic fluid. This management involves frequent antenatal visits with pre- and post-sugar monitoring for dietary and physical therapy. Secondly, rigorous monitoring will be done using Ultrasound and repeated lab tests via a dietary and physical monthly recall questionnaire.
  Interventions: Combination Product: Dietary intervention + Physical Activity + Monitoring

INTERVENTIONS:
Combination Product: Dietary intervention + Physical Activity + Monitoring — Dietary modifications will follow an 1800-kilocalorie structured plan that includes breakfast, two snacks, lunch, and dinner. The plan will focus on low carbohydrate intake with restrictions on lean options. Adherence will be closely monitored, with a monthly adherence questionnaire (PDAQ) to ensure tight blood sugar control.
  In terms of physical activity, a structured exercise plan will incorporate household activities, occupational tasks, and various levels of exercise, ranging from light to moderate and intense.
  Strict monitoring and follow-up will be conducted monthly using the Physical Activity Adherence Questionnaire (PAAQ). Secondly, short acting and long acting insulin dose and frquency will be monitored.
  Arms: Intensive Management Group
Other: Usual care — General advice and recommendations for a low glycemic diet include a flexible and adjusted daily calorie intake, structured meals without a fixed menu. Patients should be educated about healthy choices and empowered to manage their own health.
  Exercise recommendations should be tailored to the participant's activity level, with routine ANC counseling and no standard follow-up process.
  If lifestyle modifications are ineffective in controlling glycemic levels, glucophage and human insulin R will be prescribed.
  Arms: Conventional Management Group

SUMMARY:
This study involved two management protocols to manage diabetes in pregnancy. Sixty patients having GDM will be recruited on the basis of the OGTT and randomly allocated to two management groups. One group of patients will receive counselling and the conventional method of management. while the other group will receive a tailored diet plan and physical activity with low caloric and moderate intense exercises. Both groups will receive a dietary plan based on their sugar levels weekly basis and physical activity with pharmacotherapy to adjust their sugar levels, while the intensive group will have rigorous monitoring on a monthly basis and frequent visits with repeated lab checks. This will help us to reduce short and long-term complications with improved maternal and neonatal outcomes.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy of conventional versus intensive management strategies for Gestational Diabetes Mellitus (GDM) and their impact on maternal and fetal outcomes. The study will enrol 60 pregnant women diagnosed with GDM at 24-28 weeks of gestation. Participants will be randomly assigned to either a conventional group, which receives standard monthly follow-up and counselling, or an intensive group, which receives proactive weekly monitoring, personalised diet and exercise plans, and stricter glycemic targets. The primary outcomes include differences in glycemic control (glucose, HbA1c), levels of the biomarker CMPF, and the incidence of maternal and neonatal complications. Data will be collected throughout pregnancy and postpartum, and analyzed using statistical methods in SPSS to determine the superior management approach for improving health outcomes in GDM.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 18-45 years
* Gestational age at enrollment 24 - 28 weeks
* Patients having Hba1c levels less then 6%

Exclusion Criteria:

* Patients having twin pregnancies
* Patients having PCOS
* Diabetes diagnosed prior to pregnancy
* Patients having severe hypertension
* Patients having renal diseases
* Patients using glucose altering medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c Levels | Baseline (24-28 weeks), Late Pregnancy/Delivery (37-38 weeks), Postpartum (42-45 weeks)
  HbA1c is measured using high-performance liquid chromatography (HPLC). Values will be compared from baseline to delivery/late pregnancy and postpartum to assess improvement or deterioration in glycemic control.
Physical Activity Level (PAQ) | Conventional Management: Baseline, Delivery (37-38 weeks), Postpartum (42-45 weeks) Intensive Management: Baseline, 2nd Visit (32-34 weeks), 3rd Visit (36-38 weeks), 4th Visit (40-42 weeks), Postpartum (42-45 weeks)
  Physical activity is assessed using the Physical Activity Questionnaire (PAQ), an ordinal scale ranging from 1 to 5. A score ≤2 indicates sedentary activity, while a score ≥3 indicates active physical activity levels. Higher scores reflect greater physical activity engagement.

SECONDARY OUTCOMES:
Fasting or Random Blood Glucose Levels | Baseline; Delivery; 6-12 weeks postpartum
  Blood glucose is measured using the enzymatic glucose oxidase method. A fasting value ≥92 mg/dL is considered abnormal, and a random value ≥200 mg/dL suggests hyperglycemia.
Serum Insulin Levels | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  Insulin is measured using chemiluminescent immunoassay. A fasting insulin level >25 μIU/mL indicates hyperinsulinemia.
Serum CMPF | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  Serum CMPF quantified using ELISA or mass spectrometry. Reported as a continuous variable; higher values indicate increased furan fatty acid levels.
Total Cholesterol | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  Total cholesterol measured using enzymatic colorimetric assay; interpreted according to pregnancy-adjusted reference ranges.
LDL Cholesterol | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  LDL measured directly or calculated using Friedewald formula; optimal levels <100 mg/dL.
HDL Cholesterol | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  HDL analyzed using direct enzymatic methods; low HDL defined as <50 mg/dL in pregnancy.
Serum Creatinine | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  Serum creatinine measured using Jaffe or enzymatic assay; pregnancy reference range 0.4-0.8 mg/dL.
Complete Blood Count (CBC) | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  Includes hemoglobin, white blood cells, and platelet counts measured via automated hematology analyzer.
Amniotic Fluid Index (AFI) | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  AFI measured using obstetric ultrasound; values <8 cm indicate oligohydramnios, >25 cm polyhydramnios.
Estimated Fetal Weight (EFW) | Conventional Care Group: Baseline, Delivery. Intensive Care Group: Baseline, 32-34 weeks gestation, 36-38 weeks gestation, 40-42 weeks gestation, 6-12 weeks postpartum.
  EFW calculated using Hadlock fetal biometry formula; macrosomia defined as >4000 g.
Mode of Delivery | Delivery (37-38 weeks)
  Newborn weight measured using a calibrated digital scale. Low birth weight <2500 g; macrosomia >4000 g.
Neonatal Jaundice | Postpartum (42-45 days)
  Defined as total serum bilirubin >5 mg/dL in the first 24 hours or above age-specific nomogram.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kausar Tayyab, PhD*, Principal Investigator — Institute of Basic Medical Sciences, Khyber Medical University; Dr Rubina Nazli, PhD, Principal Investigator — Institute of Basic Medical Sciences, Khyber Medical University; Dr Arshad Hussain, PhD, Principal Investigator — Northwest General Hospital, Peshawar; Dr Ehtesham, PhD, Principal Investigator — Institute of Basic Medical Sciences, Khyber Medical University
Locations (2):
- Pakistan (2):
  - Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa
  - Northwest General Hospital, Peshawar, Khyber Pakhtunkhwa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications from this study will be made available to qualified researchers for legitimate scientific research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 12 months after the publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal approved by the study's principal investigator and the Institutional Review Board (IRB) of Khyber Medical University. Proposals should be directed to the corresponding author. Data will be shared via a secure, password-protected platform after signing a data use agreement.

REFERENCES:
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Wang H, Li N, Chivese T, Werfalli M, Sun H, Yuen L, Hoegfeldt CA, Elise Powe C, Immanuel J, Karuranga S, Divakar H, Levitt N, Li C, Simmons D, Yang X; IDF Diabetes Atlas Committee Hyperglycaemia in Pregnancy Special Interest Group. IDF Diabetes Atlas: Estimation of Global and Regional Gestational Diabetes Mellitus Prevalence for 2021 by International Association of Diabetes in Pregnancy Study Group's Criteria. Diabetes Res Clin Pract. 2022 Jan;183:109050. doi: 10.1016/j.diabres.2021.109050. Epub 2021 Dec 6. PMID 34883186
- [Background] Prentice KJ, Luu L, Allister EM, Liu Y, Jun LS, Sloop KW, Hardy AB, Wei L, Jia W, Fantus IG, Sweet DH, Sweeney G, Retnakaran R, Dai FF, Wheeler MB. The furan fatty acid metabolite CMPF is elevated in diabetes and induces beta cell dysfunction. Cell Metab. 2014 Apr 1;19(4):653-66. doi: 10.1016/j.cmet.2014.03.008. PMID 24703697
- [Background] American Diabetes Association Professional Practice Committee. 15. Management of Diabetes in Pregnancy: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S282-S294. doi: 10.2337/dc24-S015. PMID 38078583
- [Background] Asaad G, Soria-Contreras DC, Bell RC, Chan CB. Effectiveness of a Lifestyle Intervention in Patients with Type 2 Diabetes: The Physical Activity and Nutrition for Diabetes in Alberta (PANDA) Trial. Healthcare (Basel). 2016 Sep 27;4(4):73. doi: 10.3390/healthcare4040073. PMID 27690122
- [Background] Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004 Oct;36(10):1750-60. doi: 10.1249/01.mss.0000142303.49306.0d. PMID 15595297